CLINICAL TRIAL: NCT02090413
Title: A Phase 4, Randomized, Double-Blind Study With a Safety Extension Period to Evaluate the Effect of Aspirin on Flushing Events in Subjects With Relapsing-Remitting Multiple Sclerosis Treated With Tecfidera® (Dimethyl Fumarate) Delayed-Release Capsules
Brief Title: Phase 4 Study of Effect of Aspirin on Flushing in Dimethyl Fumarate-Treated Participants With Relapsing-Remitting Multiple Sclerosis
Acronym: ASSURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109MS406; 2013-001895-40 (EudraCT Number)
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: multiple sclerosis; flushing; aspirin
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Flushing | interventions — Dimethyl Fumarate; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DMF + ASA 150 mg BID (Experimental): DMF 120 mg taken BID for the first 7 days and 240 mg BID from Week 2 through Week 48.
  ASA 150 mg is taken BID from Day 1 through Week 4. (Between Weeks 5 and 8, ASA is prohibited; between Weeks 9 and 48, ASA is allowed as needed.)
  Interventions: Drug: dimethyl fumarate; Drug: acetylsalicylic acid
- DMF + ASA 75 mg QAM (Experimental): DMF 120 mg taken BID for the first 7 days and 240 mg BID from Week 2 through Week 48.
  ASA 75 mg is taken in the morning (QAM) and ASA-Placebo is taken in the evening (QPM) from Day 1 through Week 4. (Between Weeks 5 and 8, ASA is prohibited; between Weeks 9 and 48, ASA is allowed as needed.)
  Interventions: Drug: dimethyl fumarate; Drug: acetylsalicylic acid; Drug: ASA-Placebo
- DMF + ASA-Placebo BID (Experimental): DMF 120 mg taken BID for the first 7 days and 240 mg BID from Week 2 through Week 48.
  ASA-Placebo is taken BID from Day 1 through Week 4. (Between Weeks 5 and 8, ASA is prohibited; between Weeks 9 and 48, ASA is allowed as needed.)
  Interventions: Drug: dimethyl fumarate; Drug: ASA-Placebo

INTERVENTIONS:
Drug: dimethyl fumarate
  Other Names: BG00012; Tecfidera; DMF
Drug: acetylsalicylic acid — enteric-coated capsule
  Other Names: ASA; aspirin
  Arms: DMF + ASA 150 mg BID; DMF + ASA 75 mg QAM
Drug: ASA-Placebo — matched placebo
  Other Names: placebo
  Arms: DMF + ASA 75 mg QAM; DMF + ASA-Placebo BID

SUMMARY:
The primary objective of the study is to evaluate whether 150 mg enteric-coated aspirin (acetylsalicylic acid [ASA]) taken twice a day (BID) with dimethyl fumarate (DMF) administration or 75 mg enteric-coated ASA taken once daily in the morning (QAM) with DMF administration reduces the incidence and/or severity of flushing events in subjects with relapsing-remitting multiple sclerosis (RRMS) compared with ASA-placebo administered with DMF in the clinical practice setting.

Secondary objectives of this study are: to evaluate the safety and tolerability of DMF administered with and without enteric-coated ASA in the clinical practice setting; to evaluate the impact of DMF administration on quality of life as measured by the Short Form 36 (SF-36®) and European Quality of Life - 5 Dimensions - 5 Levels (EQ-5D-5L) questionnaires.

ELIGIBILITY:
Key Inclusion Criteria:

* Naïve to fumaric acid esters (e.g. DMF, Fumaderm, compounded fumarates)
* Diagnosed with RRMS and satisfies the approved therapeutic indication for DMF
* Participants of childbearing potential must practice effective contraception and be willing and able to continue contraception throughout the study
* Ability to complete the tolerability scales accurately using the electronic diary (eDiary) and ability to complete the paper Flushing Diaries

Key Exclusion Criteria:

* Inability or unwillingness to comply with study requirements or, at the discretion of the Investigator, is deemed unsuitable for study participation
* One or more major comorbidities that, in the opinion of the Investigator, may affect the outcome of the study or otherwise makes the subject an unsuitable candidate for study participation. The prevailing product labels for both DMF and ASA should be used as guides
* Known active malignancies (subjects with cutaneous basal cell carcinoma that has been completely excised prior to study entry remain eligible)
* Chronic use (≥7 consecutive days) of ASA- or nonsteroidal anti-inflammatory drugs (NSAID)-containing products within the month prior to enrollment in the study
* A known intolerance to ASA
* Active peptic ulceration or a history of peptic ulceration, hemophilia or other clotting disorders, or gout
* Known hypersensitivity reactions (e.g., bronchospasm, rhinitis, urticaria) in response to ASA or NSAID administration
* Impaired hepatic or renal function, in the opinion of the investigator
* Female subject is pregnant, lactating, or will be attempting to become pregnant during the Double-Blind Period (first 12 weeks) of the study
* Currently participating in another interventional clinical trial

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (17):
- Ireland (2):
  - Research Site, Cork
  - Research Site, Dublin
- United Kingdom (15):
  - Research Site, Basingstoke
  - Research Site, Birmingham
  - Research Site, Cardiff
  - Research Site, Edinburgh
  - Research Site, Exeter
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Plymouth
  - Research Site, Salford
  - Research Site, Swansea

RESULTS

PARTICIPANT FLOW:
Groups:
- DMF + ASA-Placebo BID: Dimethyl fumarate (DMF) 120 mg taken twice daily (BID) for the first 7 days and 240 mg BID from Week 2 through Week 48. Acetylsalicylic acid (ASA)-Placebo taken BID from Day 1 through Week 4. (Between Weeks 5 and 8, ASA was prohibited; between Weeks 9 and 48, ASA was allowed as needed.)
- DMF + ASA 75 mg QAM: DMF 120 mg BID for the first 7 days and 240 mg BID from Week 2 through Week 48. ASA 75 mg QAM and ASA-Placebo in the evening from Day 1 through Week 4. (Between Weeks 5 and 8, ASA was prohibited; between Weeks 9 and 48, ASA was allowed as needed.)
- DMF + ASA 150 mg BID: DMF 120 mg BID for the first 7 days and 240 mg BID from Week 2 through Week 48. ASA 150 mg BID from Day 1 through Week 4. (Between Weeks 5 and 8, ASA was prohibited; between Weeks 9 and 48, ASA was allowed as needed.)
Period: Overall Study
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Started | 81 | 80 | 80
Completed | 62 | 60 | 57
Not Completed | 19 | 20 | 23
Not completed — Adverse Event | 11 | 15 | 20
Not completed — Flushing event | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Investigator Decision | 1 | 1 | 0
Not completed — Other | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- DMF + ASA-Placebo BID: DMF 120 mg taken BID for the first 7 days and 240 mg BID from Week 2 through Week 48. ASA-Placebo taken BID from Day 1 through Week 4. (Between Weeks 5 and 8, ASA was prohibited; between Weeks 9 and 48, ASA was allowed as needed.)
- Total: Total of all reporting groups
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID | Total
Number analyzed (Participants) | 81 | 80 | 80 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.17 (10.63) | 39.48 (8.48) | 40.16 (8.23) | 39.94 (9.15)
Gender [Count of Participants; unit: Participants]
  Female | 59 | 62 | 60 | 181
  Male | 22 | 18 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Overall Flushing Events During the First 4 Weeks of Treatment, as Assessed by the Modified Global Flushing Severity Scale (MGFSS)
Description: Participant-reported flushing events during the first 4 weeks treatment, recorded on the hand-held participant reporting device (eDiary) as assessed by MGFSS. The MGFSS measures the side effects related to flushing during the past 24 hours. Flushing means redness, warmth, tingling or itching of the skin. Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects). Day 1 data are not included in the analysis because MGFSS question refers to last 24 hours flushing score.
Time Frame: Day 2 to Week 4
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug); n=number of participants evaluable at given time point.
Measure: Number; unit: percentage of participants
Groups:
- DMF + ASA-Placebo BID: DMF 120 mg BID for the first 7 days and 240 mg BID from Week 2 through Week 48. ASA-Placebo BID from Day 1 through Week 4. (Between Weeks 5 and 8, ASA was prohibited; between Weeks 9 and 48, ASA was allowed as needed.)
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 80 | 79 | 80
percentage of participants
  Weeks 1-4 combined; n=80, 79, 80 | 90.0 | 92.4 | 88.8
  Week 1; n=80, 77, 80 | 83.8 | 85.7 | 83.8
  Week 2; n=77, 76, 79 | 76.6 | 61.8 | 69.6
  Week 3; n=74, 74, 76 | 73.0 | 55.4 | 53.9
  Week 4; n=72, 71, 71 | 59.7 | 54.9 | 54.9
Statistical Analysis 1: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Weeks 1-4 combined; Test type: Superiority or Other; Difference in percentage = 2.4, 95% CI 2-sided [-6.4 to 11.2] — Two sided 95% CI of difference in proportions was constructed based on the normal approximation to the binomial distribution
Statistical Analysis 2: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Weeks 1-4 combined; Test type: Superiority or Other; Difference in percentage = -1.3, 95% CI 2-sided [-10.8 to 8.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Week 1; Test type: Superiority or Other; Difference in percentage = 2.0, 95% CI 2-sided [-9.3 to 13.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Week 1; Test type: Superiority or Other; Difference in percentage = 0.0, 95% CI 2-sided [-11.4 to 11.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Week 2; Test type: Superiority or Other; Difference in percentage = -14.8, 95% CI 2-sided [-29.2 to -0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Week 2; Test type: Superiority or Other; Difference in percentage = -7.0, 95% CI 2-sided [-20.9 to 6.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Week 3; Test type: Superiority or Other; Difference in percentage = -17.6, 95% CI 2-sided [-32.8 to -2.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Week 3; Test type: Superiority or Other; Difference in percentage = -19.0, 95% CI 2-sided [-34.1 to -3.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Week 4; Test type: Superiority or Other; Difference in percentage = -4.8, 95% CI 2-sided [-21.0 to 11.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Week 4; Test type: Superiority or Other; Difference in percentage = -4.8, 95% CI 2-sided [-21.0 to 11.4] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Participants Reporting Overall Flushing Events During the First 4 Weeks of Treatment, as Assessed by the Modified Flushing Severity Scale (MFSS)
Description: Participant-reported flushing events during the first 4 weeks of treatment recorded on the eDiary as assessed by MFSS. MFSS questionnaire measures the side effects related to flushing following drug administration. Flushing means redness, warmth, tingling or itching of the skin. This questionnaire relates only to the period of time since the investigational drug was administered and was to be completed within 10 hours of taking the study drug (2 times/day). Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Day 1 to Week 4
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug).
Measure: Number; unit: percentage of participants
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 80 | 78 | 80
percentage of participants
  Overall flushing events | 91.3 | 96.2 | 96.3
  Overall redness events | 90.0 | 88.5 | 88.8
  Overall warmth events | 92.5 | 97.4 | 97.5
  Overall tingling events | 81.3 | 87.2 | 86.3
  Overall itching events | 87.5 | 79.5 | 76.3
Statistical Analysis 1: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Overall flushing events; Test type: Superiority or Other; Difference in percentage = 4.9, 95% CI 2-sided [-2.6 to 12.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Overall flushing events; Test type: Superiority or Other; Difference in percentage = 5.0, 95% CI 2-sided [-2.5 to 12.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Overall redness events; Test type: Superiority or Other; Difference in percentage = -1.5, 95% CI 2-sided [-11.2 to 8.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Overall redness events; Test type: Superiority or Other; Difference in percentage = -1.3, 95% CI 2-sided [-10.8 to 8.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Overall warmth events; Test type: Superiority or Other; Difference in percentage = 4.9, 95% CI 2-sided [-1.8 to 11.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Overall warmth events; Test type: Superiority or Other; Difference in percentage = 5.0, 95% CI 2-sided [-1.7 to 11.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Overall tingling events; Test type: Superiority or Other; Difference in percentage = 5.9, 95% CI 2-sided [-5.4 to 17.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Overall tingling events; Test type: Superiority or Other; Difference in percentage = 5.0, 95% CI 2-sided [-6.4 to 16.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Overall itching events; Test type: Superiority or Other; Difference in percentage = -8.0, 95% CI 2-sided [-19.5 to 3.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Overall itching events; Test type: Superiority or Other; Difference in percentage = -11.3, 95% CI 2-sided [-23.1 to 0.6] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Worst Severity Scores of Overall Flushing During the First 4 Weeks of Treatment, as Assessed by MGFSS
Description: Worst severity of participant-reported flushing events during the first 4 weeks of treatment recorded on the eDiary as assessed by MGFSS. The MGFSS measures the side effects related to flushing during the past 24 hours. Flushing means redness, warmth, tingling or itching of the skin. Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects). Day 1 data are not included in the analysis because MGFSS question refers to last 24 hours flushing score.
Time Frame: Day 2 to Week 4
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 80 | 79 | 80
units on a scale | 4.36 (2.66) | 3.99 (2.63) | 3.93 (2.47)

4. Primary Outcome: Worst Severity Scores of Overall Flushing During the First 4 Weeks of Treatment, as Assessed by MFSS
Description: Worst severity of participant-reported flushing events during the first 4 weeks of treatment recorded on the eDiary as assessed by MFSS. MFSS questionnaire measures the side effects related to flushing following drug administration. Flushing means redness, warmth, tingling or itching of the skin.This questionnaire relates only to the period of time since the investigational drug was administered and was to be completed within 10 hours of taking the study drug (2 times/day). Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Day 1 to Week 4
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 80 | 78 | 80
units on a scale
  Overall flushing | 4.84 (2.77) | 4.73 (2.43) | 4.78 (2.53)
  Redness | 4.83 (2.69) | 4.65 (2.73) | 4.34 (2.67)
  Warmth | 5.03 (2.54) | 4.88 (2.38) | 4.9 (2.46)
  Tingling | 3.31 (2.38) | 3.62 (2.53) | 3.3 (2.30)
  Itching | 3.7 (2.55) | 3.64 (2.76) | 3.23 (2.66)

5. Secondary Outcome: Percentage of Participants Reporting Overall Flushing Events During Weeks 5-8 and Weeks 9-12 of Treatment, as Assessed by MGFSS
Description: Participant-reported flushing events during Weeks 5-8 and Weeks 9-12 of the study recorded on the eDiary as assessed by MGFSS. The MGFSS measures the side effects related to flushing during the past 24 hours. Flushing means redness, warmth, tingling or itching of the skin. Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Week 5 to Week 12
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug). n=number of evaluable participants at given time period.
Measure: Number; unit: percentage of participants
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 80 | 79 | 80
percentage of participants
  Weeks 5-8 combined; n=71, 71, 70 | 74.6 | 73.2 | 80.0
  Weeks 9-12 combined; n=67, 62, 65 | 61.2 | 67.7 | 76.9
Statistical Analysis 1: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = -1.4, 95% CI 2-sided [-15.8 to 13.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = 5.4, 95% CI 2-sided [-8.4 to 19.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 6.5, 95% CI 2-sided [-9.9 to 23.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 15.7, 95% CI 2-sided [0.2 to 31.3] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants Reporting Overall Flushing Events During Weeks 5-8 and Weeks 9-12 of Treatment, as Assessed by MFSS
Description: Participant-reported flushing events during Weeks 5-8 and Weeks 9-12 of the study recorded on the eDiary as assessed by MFSS. MFSS questionnaire measures the side effects related to flushing following drug administration. Flushing means redness, warmth, tingling or itching of the skin. This questionnaire relates only to the period of time since the investigational drug was administered and was to be completed within 10 hours of taking the study drug (2 times/day). Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Week 5 to Week 12
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug).
Measure: Number; unit: percentage of participants
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 80 | 78 | 80
percentage of participants
  Overall Flushing, Weeks 5-8 combined; n=71, 70, 70 | 80.3 | 82.9 | 84.3
  Overall Flushing, Weeks 9-12 combined;n=68, 65, 65 | 66.2 | 69.2 | 78.5
  Redness, Weeks 5-8 combined; n=71, 70, 70 | 77.5 | 75.7 | 81.4
  Redness, Weeks 9-12 combined; n=68, 65, 65 | 70.6 | 61.5 | 73.8
  Warmth, Weeks 5-8 combined; n=71, 70, 70 | 80.3 | 80.0 | 82.9
  Warmth, Weeks 9-12 combined; n=68, 65, 65 | 70.6 | 70.8 | 75.4
  Tingling, Weeks 5-8 combined; n=71, 70, 70 | 57.7 | 55.7 | 71.4
  Tingling, Weeks 9-12 combined; n=68, 65, 65 | 54.4 | 49.2 | 61.5
  Itching, Weeks 5-8 combined; n=71, 70, 70 | 54.9 | 64.3 | 64.3
  Itching, Weeks 9-12 combined; n=68, 65, 65 | 48.5 | 52.3 | 56.9
Statistical Analysis 1: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Overall flushing, Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = 2.6, 95% CI 2-sided [-10.2 to 15.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Overall flushing, Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = 4.0, 95% CI 2-sided [-8.6 to 16.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Overall flushing, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 3.1, 95% CI 2-sided [-12.8 to 18.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Overall flushing, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 12.3, 95% CI 2-sided [-2.8 to 27.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Redness, Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = -1.8, 95% CI 2-sided [-15.7 to 12.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Redness, Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = 4.0, 95% CI 2-sided [-9.4 to 17.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Redness, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = -9.0, 95% CI 2-sided [-25.1 to 7.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Redness, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 3.3, 95% CI 2-sided [-12.0 to 18.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Warmth, Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = -0.3, 95% CI 2-sided [-13.5 to 12.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Warmth, Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = 2.6, 95% CI 2-sided [-10.2 to 15.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Warmth, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 0.2, 95% CI 2-sided [-15.3 to 15.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Warmth, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 4.8, 95% CI 2-sided [-10.3 to 19.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Tingling, Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = -2.0, 95% CI 2-sided [-18.4 to 14.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Tingling, Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = 13.7, 95% CI 2-sided [-1.9 to 29.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Tingling, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = -5.2, 95% CI 2-sided [-22.1 to 11.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Tingling, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 7.1, 95% CI 2-sided [-9.6 to 23.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Itching, Weeks 5-8 combined; Test type: Superiority or Other; Difference in percentage = 9.4, 95% CI 2-sided [-6.8 to 25.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Itching, Weeks 5-8; Test type: Superiority or Other; Difference in percentage = 9.4, 95% CI 2-sided [-6.8 to 25.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Itching, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 3.8, 95% CI 2-sided [-13.2 to 20.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Itching, Weeks 9-12 combined; Test type: Superiority or Other; Difference in percentage = 8.4, 95% CI 2-sided [-8.5 to 25.3] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Worst Severity Scores of Overall Flushing During Weeks 5-8 and Weeks 9-12 of the Study, as Assessed by MGFSS
Description: Worst severity of participant-reported flushing events during Weeks 5-8 and Weeks 9-12 of the study recorded on the eDiary as assessed by MGFSS. The MGFSS measures the side effects related to flushing during the past 24 hours. Flushing means redness, warmth, tingling or itching of the skin. Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Week 5 to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 80 | 79 | 80
units on a scale
  Weeks 5-8 combined; n=71, 71, 70 | 3.00 (2.61) | 2.83 (2.4) | 3.47 (2.64)
  Weeks 9 to 12 combined; n=67, 62, 65 | 2.43 (2.72) | 2.81 (2.76) | 2.95 (2.5)

8. Secondary Outcome: Worst Severity Scores of Overall Flushing During Weeks 5-8 and Weeks 9-12 of the Study, as Assessed by MFSS
Description: Worst severity of participant-reported flushing events during Weeks 5-8 and Weeks 9-12 of the study recorded on the eDiary as assessed by MFSS. MFSS questionnaire measures the side effects related to flushing following drug administration. Flushing means redness, warmth, tingling or itching of the skin. This questionnaire relates only to the period of time since the investigational drug was administered and was to be completed within 10 hours of taking the study drug (2 times/day). Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Week 5 to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 80 | 78 | 80
units on a scale
  Overall Flushing, Weeks 5-8 combined; n=71, 70, 70 | 3.37 (2.8) | 3.24 (2.57) | 3.57 (2.45)
  Overall Flushing, Weeks 9-12 combined;n=68, 65, 65 | 2.5 (2.65) | 3.15 (2.98) | 3.45 (2.74)
  Redness, Weeks 5-8 combined; n=71, 70, 70 | 3.27 (2.9) | 2.83 (2.54) | 3.51 (2.58)
  Redness, Weeks 9-12 combined; n=68, 65, 65 | 2.57 (2.55) | 2.75 (3.13) | 3.4 (2.93)
  Warmth, Weeks 5-8 combined; n=71, 70, 70 | 3.3 (2.71) | 3.11 (2.45) | 3.49 (2.54)
  Warmth, Weeks 9-12 combined; n=68, 65, 65 | 2.66 (2.52) | 3.06 (2.97) | 3.45 (2.85)
  Tingling, Weeks 5-8 combined; n=71, 70, 70 | 2.03 (2.41) | 2.07 (2.5) | 2.79 (2.56)
  Tingling, Weeks 9-12 combined; n=68, 65, 65 | 1.71 (2.17) | 1.78 (2.43) | 2.54 (2.69)
  Itching, Weeks 5-8 combined; n=71, 70, 70 | 1.92 (2.35) | 2.17 (2.32) | 2.64 (2.59)
  Itching, Weeks 9-12 combined; n=68, 65, 65 | 1.51 (2.04) | 1.69 (2.15) | 2.17 (2.52)

9. Secondary Outcome: Duration of Flushing Episodes During Weeks 1-4, 5-8 and 9-12 of the Study, as Assessed by MGFSS
Description: Duration of participant-reported flushing events during weeks 1-4, 5-8 and 9-12 of the study recorded on the eDiary as assessed by MGFSS. The MGFSS measures the side effects related to flushing during the past 24 hours. Flushing means redness, warmth, tingling or itching of the skin. Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects).
Time Frame: Day 1 to Week 12
Population: Although designated as a secondary endpoint, the duration of flushing events based on MGFSS could not be calculated because specific flushing events with start and end times was not captured in the MGFSS.
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Duration of Flushing Episodes During Weeks 1-4, 5-8 and 9-12 of the Study, as Assessed by MFSS
Description: Duration of participant-reported flushing events during weeks 1-4, 5-8 and 9-12 of the study recorded on the eDiary as assessed by MFSS. MFSS questionnaire measures the side effects related to flushing following drug administration. Flushing means redness, warmth, tingling or itching of the skin. This questionnaire relates only to the period of time since the investigational drug was administered and was to be completed within 10 hours of taking the study drug (2 times/day). Each question is rated on a scale from 0 (no flushing side effects) to 10 (extreme flushing side effects). For participants with more than 1 flushing event during a visit interval, the average duration for the visit interval was used.
Time Frame: Day 1 to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
hours
  Weeks 1-4 combined; n=73, 75, 77 | 0.69 (0.44) | 0.8 (0.59) | 1.11 (1.16)
  Weeks 5-8 combined; n=57, 58, 59 | 1.06 (2.12) | 0.73 (0.52) | 1.08 (1.18)
  Weeks 9-12 combined; n=45, 45, 51 | 0.66 (0.52) | 0.69 (0.59) | 0.79 (0.94)
Statistical Analysis 1: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Weeks 1-4 combined; Test type: Superiority or Other; Mean Difference (Final Values) = -0.145, 95% CI 2-sided [-0.414 to 0.125] — Analysis of variance model (ANCOVA) model was used with treatment, center as effects and baseline characteristics as covariates
Statistical Analysis 2: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Weeks 1-4 combined; Test type: Superiority or Other; Mean Difference (Final Values) = -0.392, 95% CI 2-sided [-0.656 to -0.128] — ANCOVA model was used with treatment, center as effects and baseline characteristics as covariates
Statistical Analysis 3: Comparison: DMF + ASA 75 mg QAM vs DMF + ASA 150 mg BID; Weeks 1-4 combined; Test type: Superiority or Other; Mean Difference (Final Values) = -0.247, 95% CI 2-sided [-0.507 to 0.012] — ANCOVA model was used with treatment, center as effects and baseline characteristics as covariates
Statistical Analysis 4: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Weeks 5-8 combined; Test type: Superiority or Other; Mean Difference (Final Values) = 0.376, 95% CI 2-sided [-0.193 to 0.945] — ANCOVA model was used with treatment, center as effects and baseline characteristics as covariates
Statistical Analysis 5: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Weeks 5-8 combined; Test type: Superiority or Other; Mean Difference (Final Values) = 0.069, 95% CI 2-sided [-0.498 to 0.635] — ANCOVA model was used with treatment, center as effects and baseline characteristics as covariates
Statistical Analysis 6: Comparison: DMF + ASA 75 mg QAM vs DMF + ASA 150 mg BID; Weeks 5-8 combined; Test type: Superiority or Other; Mean Difference (Final Values) = -0.308, 95% CI 2-sided [-0.867 to 0.251] — ANCOVA model was used with treatment, center as effects and baseline characteristics as covariates
Statistical Analysis 7: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 75 mg QAM; Weeks 9-12 combined; Test type: Superiority or Other; Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.308 to 0.355] — ANCOVA model was used with treatment, center as effects and baseline characteristics as covariates
Statistical Analysis 8: Comparison: DMF + ASA-Placebo BID vs DMF + ASA 150 mg BID; Weeks 9-12 combined; Test type: Superiority or Other; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.374 to 0.254] — ANCOVA model was used with treatment, center as effects and baseline characteristics as covariates
Statistical Analysis 9: Comparison: DMF + ASA 75 mg QAM vs DMF + ASA 150 mg BID; Weeks 9-12 combined; Test type: Superiority or Other; Mean Difference (Final Values) = -0.084, 95% CI 2-sided [-0.4 to 0.232] — ANCOVA model was used with treatment, center as effects and baseline characteristics as covariates

11. Secondary Outcome: Number of Participants With Self-Reported Flushing Events During Weeks 13 to 48
Description: Participant-reported flushing events (which include redness, warmth, tingling, and/or itching of the skin) during Weeks 13 to 48 of treatment were recorded in the CRF.
Time Frame: Week 13 to Week 48
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug).
Measure: Number; unit: participants
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
participants | 36 | 35 | 42

12. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events (AEs), Serious AEs (SAEs), and Discontinuations Due to AEs in the First 12 Weeks
Description: AE: any untoward medical occurrence that does not necessarily have a causal relationship with treatment. SAE: any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity, or; results in a congenital anomaly/birth defect. An SAE may also be any other medically important event that, in the opinion of the Investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed above. A treatment-emergent AE is defined as any AE that occurs after the first administration of DMF or ASA/Placebo drug.
Time Frame: Day 1 to Week 12
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug).
Measure: Number; unit: participants
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
participants
  Any event | 66 | 68 | 63
  Moderate or severe event | 24 | 38 | 26
  Severe event | 3 | 5 | 8
  Related event | 35 | 38 | 40
  Serious event | 1 | 1 | 2
  Discontinued treatment due to event | 5 | 9 | 12
  Discontinued study due to event | 5 | 9 | 13

13. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent AEs, SAEs, and Discontinuations Due to AEs in Weeks 13 to 48
Description: as for outcome 12
Time Frame: Week 13 to Week 48
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug).
Measure: Number; unit: participants
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
participants
  Any event | 66 | 68 | 66
  Moderate or severe event | 40 | 50 | 51
  Severe event | 5 | 12 | 12
  Related event | 45 | 42 | 49
  Serious event | 3 | 7 | 3
  Discontinued treatment due to event | 9 | 6 | 10
  Discontinued study due to event | 9 | 6 | 10

14. Secondary Outcome: Number of Participants Discontinuing Treatment and Discontinuing the Study Due to Treatment-emergent Flushing AEs in the First 12 Weeks
Description: A treatment-emergent AE is defined as any AE that occurs after the first administration of DMF or ASA/Placebo drug. Flushing AEs include redness, warmth, tingling, and/or itching of the skin.
Time Frame: Day 1 to Week 12
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug).
Measure: Number; unit: participants
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
participants
  Discontinuing treatment | 0 | 0 | 2
  Discontinuing study | 0 | 0 | 2

15. Secondary Outcome: Number of Participants Discontinuing Treatment and Discontinuing the Study Due to Treatment-Emergent Flushing AEs in Weeks 13 to 48
Description: as for outcome 14
Time Frame: Week 13 to Week 48
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug).
Measure: Number; unit: participants
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
participants
  Discontinuing treatment | 2 | 0 | 0
  Discontinuing study | 2 | 0 | 0

16. Secondary Outcome: Change From Baseline at Weeks 24 and 48 in Quality of Life Measurements as Assessed by Short Form-36 (SF-36) Questionnaire: Physical Component Summary (PCS)
Description: SF-36 is a self-administered, generic health status questionnaire consisting of 36 questions that measure 8 health concepts: physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems and mental health. The score for a domain is an average of the individual question scores, which are scaled 0 (worst health-related quality of life) to 100 (best health-related quality of life). Score from physical function, role physical, bodily pain, and general health domains were averaged to calculate PCS. Total score range for PCS was 0 (lowest level of physical functioning) to 100 (highest level of physical functioning).
Time Frame: Baseline, Week 24, Week 48 or early termination (ET)
Population: Evaluable participants in the Safety Population (randomized participants who received at least 1 dose of study drug); n=number of participants with an assessment at given timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
units on a scale
  Baseline; n=81, 80, 80 | 44.627 (10.822) | 41.99 (10.966) | 43.16 (11.438)
  Change at Week 24; n=68, 63, 61 | -0.014 (9.154) | 0.551 (8.473) | -1.471 (7.754)
  Change at Week 48/ET; n=68, 65, 64 | -1.008 (10.31) | -1.449 (10.964) | -2.989 (14.22)

17. Secondary Outcome: Change From Baseline at Weeks 24 and 48 in Quality of Life Measurements as Assessed by Short Form-36 (SF-36) Questionnaire: Mental Component Summary (MCS)
Description: SF-36 is a self-administered, generic health status questionnaire consisting of 36 questions that measure 8 health concepts: physical functioning, role limitations due to physical problems, bodily pain, general health perception, vitality, social functioning, role limitations due to emotional problems and mental health. The score for a domain is an average of the individual question scores, which are scaled 0 (worst health-related quality of life) to 100 (best health-related quality of life). Score from mental health, role emotional, social functioning, and vitality domains were averaged to calculate MCS. Total score range for MCS was 0 (lowest level of physical functioning) to 100 (highest level of physical functioning).
Time Frame: Baseline, Week 24, Week 48 or ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
units on a scale
  Baseline; n=81, 80, 80 | 47.413 (8.772) | 45.048 (10.531) | 46.496 (10.812)
  Change at Week 24; n=68, 63, 61 | -0.139 (11.66) | -0.893 (10.059) | -0.312 (12.251)
  Change at Week 48/ET; n=68, 65, 64 | -0.976 (13.759) | -2.081 (13.733) | -2.82 (15.465)

18. Secondary Outcome: Change From Baseline to Week 24 and Week 48 in Quality of Life Measurements as Assessed by the European Quality of Life 5-Dimensions Questionnaire (EQ-5D-5L) Questionnaire: Mobility
Description: EQ-5D-5L is a standardized, subject-rated instrument for use as a measure of health outcomes. The EQ 5D-5L includes 2 components: the EQ-5D-5L descriptive system and the EQ-Visual Analog Scale (EQ-VAS). The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the participant is instructed to indicate whether he or she has "no problems" (1), "some problems" (2), or "severe problems" (3). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 24, Week 48 or ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
units on a scale
  Baseline; n=81, 79, 80 | 1.877 (0.967) | 1.785 (0.887) | 1.888 (0.928)
  Change at Week 24; n=67, 63, 60 | -0.104 (0.606) | 0.095 (1.214) | -0.05 (0.467)
  Change at Week 48/ET; n=67, 63, 63 | 0.03 (0.627) | 0.079 (1.021) | 0.095 (0.56)

19. Secondary Outcome: Change From Baseline to Week 24 and Week 48 in Quality of Life Measurements as Assessed by the EQ-5D-5L Questionnaire: Self-Care
Description: EQ-5D-5L is a standardized, subject-rated instrument for use as a measure of health outcomes. The EQ 5D-5L includes 2 components: the EQ-5D-5L descriptive system and the EQ-VAS. The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the participant is instructed to indicate whether he or she has "no problems" (1), "some problems" (2), or "severe problems" (3). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 24, Week 48 or ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
units on a scale
  Baseline; n=81, 79, 80 | 1.321 (0.668) | 1.38 (0.722) | 1.363 (0.621)
  Change at Week 24; n=67, 63, 60 | -0.045 (0.442) | -0.079 (1.182) | 0.017 (0.567)
  Change at Week 48/ET; n=67, 64, 63 | -0.045 (0.367) | -0.109 (1.143) | 0.079 (0.604)

20. Secondary Outcome: Change From Baseline to Week 24 and Week 48 in Quality of Life Measurements as Assessed by the EQ-5D-5L Questionnaire: Usual Activities
Description: as for outcome 19
Time Frame: Baseline, Week 24, Week 48 or ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
units on a scale
  Baseline; n=81, 79, 80 | 1.827 (0.891) | 1.975 (0.947) | 2.025 (0.993)
  Change at Week 24; n=67, 63, 60 | -0.06 (0.694) | 0 (1.244) | -0.017 (0.725)
  Change at Week 48/ET; n=67, 64, 63 | 0.149 (0.783) | -0.016 (1.105) | 0.063 (0.896)

21. Secondary Outcome: Change From Baseline to Week 24 and Week 48 in Quality of Life Measurements as Assessed by the EQ-5D-5L Questionnaire: Pain/Discomfort
Description: as for outcome 19
Time Frame: Baseline, Week 24, Week 48 or ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
units on a scale
  Baseline; n=81, 79, 80 | 2 (0.88) | 2.038 (0.869) | 1.975 (0.941)
  Change at Week 24; n=67, 63, 60 | -0.104 (0.699) | 0 (1.032) | 0.1 (0.573)
  Change at Week 48/ET; n=67, 64, 63 | -0.09 (0.712) | 0.078 (1.117) | -0.127 (0.707)

22. Secondary Outcome: Change From Baseline to Week 24 and Week 48 in Quality of Life Measurements as Assessed by the EQ-5D-5L Questionnaire: Anxiety/Depression
Description: as for outcome 19
Time Frame: Baseline, Week 24, Week 48 or ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
units on a scale
  Baseline; n=81, 79, 80 | 1.642 (0.763) | 1.848 (0.893) | 1.763 (0.917)
  Change at Week 24; n=67, 63, 60 | -0.06 (0.903) | -0.19 (1.293) | 0 (0.803)
  Change at Week 48/ET; n=67, 63, 63 | 0.03 (0.953) | -0.127 (1.184) | -0.032 (0.842)

23. Secondary Outcome: Change From Baseline to Week 24 and Week 48 in Quality of Life Measurements as Assessed by the EQ-VAS
Description: For the EQ-VAS, the participant was instructed to draw a line on a 20-cm vertical scale at the point that best describes his or her own health, where 0 represents the "worst imaginable health state" and 100 represents the "best imaginable health state."
Time Frame: Baseline, Week 24, Week 48 or ET
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Number analyzed (Participants) | 81 | 80 | 80
units on a scale
  Baseline; n=80, 80, 80 | 78.288 (16.442) | 69.6 (19.535) | 73.438 (16.38)
  Change at Week 24; n=66, 63, 60 | -2.318 (12.579) | -0.587 (17.24) | -2.95 (16.326)
  Change at Week 48/ET; n=66, 64, 63 | -3.061 (18.053) | -0.438 (17.834) | -1.476 (13.201)

ADVERSE EVENTS:
Time Frame: Screening through Week 48
Arm/Group | DMF + ASA-Placebo BID | DMF + ASA 75 mg QAM | DMF + ASA 150 mg BID
Serious Adverse Events (participants affected / at risk) | 4/81 | 8/80 | 5/80
Other Adverse Events (participants affected / at risk) | 77/81 | 76/80 | 76/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DMF + ASA-Placebo BID (N=81) | DMF + ASA 75 mg QAM (N=80) | DMF + ASA 150 mg BID (N=80)
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Drug intolerance (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Abasia (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DMF + ASA-Placebo BID (N=81) | DMF + ASA 75 mg QAM (N=80) | DMF + ASA 150 mg BID (N=80)
Diarrhoea (Gastrointestinal disorders) | 17 | 21 | 19
Nausea (Gastrointestinal disorders) | 12 | 16 | 23
Vomiting (Gastrointestinal disorders) | 14 | 14 | 14
Abdominal pain (Gastrointestinal disorders) | 8 | 5 | 10
Abdominal pain upper (Gastrointestinal disorders) | 9 | 10 | 7
Constipation (Gastrointestinal disorders) | 3 | 7 | 5
Abdominal distension (Gastrointestinal disorders) | 6 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 4
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 4
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 20 | 15 | 16
Urinary tract infection (Infections and infestations) | 8 | 9 | 10
Lower respiratory tract infection (Infections and infestations) | 3 | 10 | 7
Sinusitis (Infections and infestations) | 2 | 1 | 5
Candida infection (Infections and infestations) | 1 | 3 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 4
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 3 | 0
Tooth infection (Infections and infestations) | 1 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Gastric infection (Infections and infestations) | 0 | 2 | 2
Ear infection (Infections and infestations) | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 2 | 1
Infected dermal cyst (Infections and infestations) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1
Eye infection (Infections and infestations) | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0
Headache (Nervous system disorders) | 16 | 14 | 18
Multiple sclerosis relapse (Nervous system disorders) | 5 | 12 | 5
Paraesthesia (Nervous system disorders) | 5 | 7 | 5
Hypoaesthesia (Nervous system disorders) | 4 | 8 | 4
Migraine (Nervous system disorders) | 2 | 2 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 3
Dizziness (Nervous system disorders) | 3 | 2 | 4
Amnesia (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Dystonia (Nervous system disorders) | 0 | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 3
Syncope (Nervous system disorders) | 1 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1
Uhthoff's phenomenon (Nervous system disorders) | 0 | 2 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 11 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Xanthelasma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 9 | 11 | 7
Influenza like illness (General disorders) | 2 | 2 | 4
Asthenia (General disorders) | 2 | 0 | 2
Chest discomfort (General disorders) | 0 | 2 | 2
Pain (General disorders) | 0 | 2 | 1
Chills (General disorders) | 0 | 0 | 2
Feeling abnormal (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 2
Depressed mood (Psychiatric disorders) | 1 | 3 | 2
Depression (Psychiatric disorders) | 5 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 1
Anger (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 2 | 0
Menorrhagia (Reproductive system and breast disorders) | 2 | 1 | 1
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 2 | 6
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vision blurred (Eye disorders) | 2 | 2 | 2
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 3
Aspartate aminotransferase abnormal (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 2 | 1
Serum ferritin decreased (Investigations) | 1 | 1 | 0
Smear cervix abnormal (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0
Flushing (Vascular disorders) | 42 | 36 | 45
Hypertension (Vascular disorders) | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 2 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Stomach ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Impetigo (Infections and infestations) | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1 | 0
Pyuria (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sensory disturbance (Nervous system disorders) | 2 | 2 | 0
Neuralgia (Nervous system disorders) | 1 | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Aphonia (Nervous system disorders) | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1
Pain (Nervous system disorders) | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail hypertrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritis generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 5 | 5
Platelet count decreased (Investigations) | 2 | 1 | 0
Blood iron decreased (Investigations) | 1 | 1 | 0
Lymphocyte count abnormal (Investigations) | 2 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood folate decreased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Vitamin B12 decreased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 3
Adverse drug reaction (General disorders) | 1 | 1 | 0
Device failure (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 1
Eye pain (Eye disorders) | 2 | 0 | 1
Colour blindness acquired (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Scleritis (Eye disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 1
Anisomastia (Reproductive system and breast disorders) | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 1 | 0
Cow's milk intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Disturbance in attention (Psychiatric disorders) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.